| $\hat{}$ | | | ICI | | E: |
|----------|---|---|-----|---|--------|
| | - | - | | | <br>ь. |
| _ | | | • | _ | . 🗕 . |

A Phase 1/Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of a Single Intraoperative Administration of CA-008 in Subjects Undergoing Unilateral Transpositional First Metatarsal Osteotomy for the Correction of Hallux Valgus Deformity

## **NCT NUMBER:**

NCT03307837

#### **DOCUMENT DATE:**

31 Mar 2018



#### STATISTICAL ANALYSIS PLAN

A Phase 1/Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of a Single Intraoperative Administration of CA-008 in Subjects Undergoing Unilateral Transpositional First Metatarsal Osteotomy for the Correction of Hallux Valgus Deformity

Protocol Number: CA-PS-2017-101

Protocol Version 3.0 Amendment 2 (30JAN2018)

SPONSORED BY

Concentric Analgesics, Inc.

PREPARED BY
Lotus Clinical Research®, LLC
100 W California Blvd, Unit 25
Pasadena, CA 91105
626-397-2390 office
info@LotusCR.com
www.LotusCR.com

This document is confidential and proprietary to **Concentric Analgesics, Inc.** Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of **Concentric Analgesics, Inc.**, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-2017-101

Statistical Analysis Plan

Date: 31Mar2018

# **DOCUMENT VERSION CONTROL**

| Version Number | Date | Comments/Changes |
|----------------|-----------|------------------|
| V1.0 | 26FEB2018 | Final SAP |


Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-2017-101

Statistical Analysis Plan Date: 31Mar2018

#### **APPROVALS**

Author:

DocuSigned by:

Signer Name: Song Liou
Signing Reason: I am the author of this document
Signing Time: 4/2/2018 9:23:57 AM PDT

85C80776CFA1404FB9C34B43BB0AA100

02-Apr-18

Thomas Graves / Song Liou

Date:

Biostatistician

Lotus Clinical Research®, LLC

Reviewed:

DocuSigned by:

| Jennifer Hesser
| Signer Name: Jennifer Nezzer
| Signing Reason: I have reviewed this document
| Signing Time: 4/2/2018 7:10:16 PM PDT
| F51546CD923C410C87CAB1F62D450C79

02-Apr-18

Date:

Jennifer Nezzer

Director, Biometrics

Lotus Clinical Research®, LLC

Approved:



05-Apr-18

Rob Allen, MD

Chief Medical Officer

Concentric Analgesics, Inc.

Date:

CONFIDENTIAL


# **TABLE OF CONTENTS**

| LIST C | OF IN-TEXT TABLES AND FIGURES | 6 |
|--------|---------------------------------------------------|----|
| LIST | OF ABBREVIATIONS (COMMONLY USED) | 7 |
| 1 | PURPOSE OF THE ANALYSES | 9 |
| 2 | PROTOCOL SUMMARY | 9 |
| 2.1 | Study Objectives | 9 |
| 2.1.1 | Primary Objectives | 9 |
| 2.1.2 | Secondary Objective | 9 |
| 2.2 | Overall Study Design and Plan | 9 |
| 2.2.1 | Study Population | 12 |
| 2.2.2 | Treatment Regimens | 12 |
| 2.2.3 | Treatment Group Assignments or Randomization | |
| 2.2.4 | Sample Size Determination | 13 |
| 3 | GENERAL ANALYSIS AND REPORTING CONVENTIONS | 13 |
| 4 | SUBJECT POPULATIONS | 14 |
| 4.1 | Analysis Populations | 14 |
| 4.2 | Disposition of Subjects | 15 |
| 4.3 | Protocol Deviations | 15 |
| 5 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 15 |
| 5.1 | Demographics and Baseline Characteristics | 15 |
| 5.2 | Medical/Surgical History | 16 |
| 5.3 | Prior and Concomitant Medications | 16 |
| 6 | MEASUREMENTS OF TREATMENT EXPOSURE and COMPLIANCE | 16 |
| 7 | EFFICACY EVALUATION | 18 |
| 7.1 | Handling of Dropouts or Missing Data | 18 |
| 7.2 | Assessment Time Windows | 18 |
| 7.3 | Exploratory Efficacy Endpoints | 18 |
| 7.4 | Analysis Methods | 19 |
| 7.4.1 | AUC Outcomes | 19 |

| 7.4.2 | Average Daily NPRS score of 2 daily diary assessments | . 19 |
|---|---|---|
| 7.4.3 | Total daily opioid consumption (in oral morphine equivalents) | . 20 |
| 7.4.4 | Proportion of patients who drop out of the study due to inadequate analgesia from Day 1 to 15. | . 21 |
| 7.4.5 | Brief Pain Inventory-short form (BPI-SF) | . 21 |
| 7.4.6 | PGE and IGE | . 21 |
| 7.4.7 | Time to First Use of Rescue Medication | . 22 |
| 7.4.8 | Percent of Subjects Taking Rescue / Use of Rescue Medication over Time | . 22 |
| 8 | SAFETY EVALUATION | . 22 |
| 8.1 | Overview of Safety Analysis Methods | . 22 |
| 8.2 | Adverse Events | . 23 |
| 8.3 | Clinical Laboratory Evaluation | . 25 |
| 8.4 | Vital Signs | . 25 |
| 8.5 | Physical Examination | . 25 |
| 8.6 | Surgical Site Assessment | . 25 |
| 8.7 | Neurosensory Assessment | . 25 |
| 8.8 | ECG Examinations | . 25 |
| 8.9 | Drugs of Abuse and Alcohol Screens, Pregnancy Test | . 25 |
| 8.10 | Patient Pain Assessment Training and Surgery Details | . 26 |
| 9 | PHARMACOKINETIC EVALUATION | . 26 |
| 10 | OTHER ANALYSES | . 27 |
| 11 | INTERIM ANALYSES AND DATA MONITORING | . 27 |
| 12 | CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL | . 27 |
| 13 | REFERENCES | . 27 |
| 14 | APPENDICES | . 28 |
| 14.1 | Tables, Figures and Listings for Final Study Report | . 28 |
| 14.1.1 | Tables | . 28 |
| 14.1.2 | Figures | . 30 |
| 14.1.3 | Listings | . 30 |

Sponsor: Concentric Analgesics, Inc. Protocol Number: CA-PS-2017-101

Statistical Analysis Plan

Date: 31Mar2018

# **LIST OF IN-TEXT TABLES AND FIGURES**

| Table 2-1 | Protocol-Specified Visits and Visit Windows | 12 |
|-----------|------------------------------------------------------|----|
| Table 7-1 | Table of Morphine Milligram Equivalents | 20 |
| Table 8-1 | Table of Imputation Rules for Missing AE Start Dates | 24 |


## LIST OF ABBREVIATIONS (COMMONLY USED)

ADaM Analysis Data Model

AE Adverse Event

ANCOVA Analysis of covariance

ANOVA Analysis of variance

ASA American Society Of Anesthesiologists

ATC Anatomical Therapeutic Chemical

AUC Area Under the Curve

BMI Body Mass Index

BP Blood Pressure

BPI-SF Brief Pain Inventory – Short Form

CDER Center for Drug Evaluation and Research

CMH Cochran Mantel Haenszel Test

CRF Case Report Form

CSR Clinical Study Report

DMC Data Monitoring Committee

ECG Electrocardiogram

EOS End of Study

ET Early Termination

FDA Food and Drug Administration

ICF Informed Consent Form

ICH International Conference on Harmonization

IGE Investigator Global Evaluation

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

MEQ morphine milligram equivalents

MMRM Mixed Model for Repeated Measures

NPRS Numerical Pain Rating Scale


PE Physical Exam

PGE Patient Global Evaluation

PK Pharmacokinetic
PT Preferred Term

SAE Serious Adverse Event/Experience

SAP Statistical Analysis Plan

SD Standard Deviation

SDTM Standard Data Table Model

SOC System Organ Class

TEAE Treatment Emergent Adverse Event

TFLs Tables, Figures and Listings

UDS Urine Drug Screen

WHO World Health Organization

WOCF Worst Observation Carried Forward


#### 1 PURPOSE OF THE ANALYSES

This statistical analysis plan (SAP) is based on protocol number CA-PS-2017-101 Version 3.0 Amendment 2 (30JAN2018) from Concentric Analgesics, Inc. The SAP will be signed off before the final database lock. The SAP contains detailed information to aid in the performance of the statistical analysis and reporting of the study data for use in the final clinical study report (CSR). This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonization (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials, the most recent ICH E3 Guideline and the Guidance for Industry: Structure and Content of Clinical Study and the most recent FDA draft Guidance for Industry - Analgesic Indications: Developing Drug and Biological Products, dated February 2014.

This SAP describes the data that will be analyzed and the subject characteristics, safety, and efficacy assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. If additional analyses are performed after database lock and unblinding to supplement the planned analyses described in this SAP, they will be clearly identified as post-hoc in the CSR.

#### 2 PROTOCOL SUMMARY

# 2.1 Study Objectives

#### 2.1.1 Primary Objectives

- To evaluate the safety and tolerability of a single intraoperative administration of CA-008 in subjects undergoing bunionectomy.
- To evaluate the pharmacokinetics of a single intraoperative administration of CA-008.

## 2.1.2 Secondary Objective

 To evaluate the efficacy of CA-008 in the management of acute postoperative pain in subjects undergoing bunionectomy.

## 2.2 Overall Study Design and Plan

This is a single-center, randomized, double-blind, placebo-controlled, single ascending dose, sequential-group Phase 1 study in subjects undergoing bunionectomy. This trial is designed to determine the recommended dose and define the toxicity profile of CA-008.

The study will be conducted utilizing an escalating dose cohort design, with sequential groups of 8 subjects each. Within each dose cohort, 6 subjects will be randomized to active, and 2 will be randomized to placebo. The initial cohort will receive the lowest planned dose of CA-008 in a fixed


Sponsor: Concentric Analgesics, Inc.

Statistical Analysis Plan Protocol Number: CA-PS-2017-101 Date: 31Mar2018

volume of administration, and will employ sentinel dosing, whereby the first 4 subjects in the first cohort will be dosed initially, before the remaining 4 subjects are dosed. If the available safety assessments for the first 4 subjects are acceptable through the first 24 hours, then the second group of 4 subjects will be dosed. Subsequent cohorts will not include sentinel dosing. There will be at least a 6-day period between cohorts, to ensure a minimum of 3 days to review safety data from the last subject in a cohort and to allow the meeting of the Data Monitoring Committee (DMC) to review the safety data from the entire cohort prior to making a decision for dose escalation. Dose escalation, or continuation of dosing, will not occur if subjects in a cohort experience intolerable treatment related AEs on active drug, as defined in the protocol.

Subjects will be screened for participation at the study site in the United States within 28 days of surgery/study drug administration. The following screening assessments will be completed: informed consent, inclusion / exclusion, demographics, medical and surgical history, prior/current medications, physical exam (PE), x-ray of surgical site, neurosensory exam of the foot / great toe (bilateral), clinical laboratory tests (chemistry/coagulation, hematology, and urinalysis), urine drug screening (UDS), alcohol breath test, serum pregnancy test, surgical site assessment, vital signs (resting blood pressure, resting pulse, oral temperature and resting respiration rate), 12-lead electrocardiograms (ECGs), subject pain assessment training, and adverse event (AE) assessment.

Subjects who meet the selection criteria at the Screening Visit and are eligible to participate in the study will be required to return to the study center within 28 days of screening. At that time, the screening assessments will again be performed (minus the x-ray and ECG) to confirm continued eligibility, and a blood draw for PK analysis will be collected. If eligible, the subject will then be randomized to treatment.

Subjects will then undergo surgery. During surgery, a total of 10 mL (for Cohorts 1-4) or 14 mL (for Cohort 5) of the investigative product will be administered into the surgical site in two applications. At time of closure of capsule, infiltration of deep soft tissue and capsule with a total of 6 mL (for Cohorts 1-4) or 9 mL (for Cohort 5) volume and instillation at cut bone with a total of 2 mL volume will be done. Then, following closure of the capsule and prior to closure of the skin and subcutaneous layer, the wound will be instilled for Cohorts 1- 4 with 2 mL volume (study drug is applied to all exposed surfaces prior to subcutaneous and skin closure) and for Cohort 5 with 2 mL of study drug will be instilled into the space under closed capsule and 1 mL of study drug applied to all exposed surfaces prior to subcutaneous and skin closure.

Time 0 will be defined as the time of completion of study drug administration. After the surgery, subjects will be monitored for 48 hours at the trial site. Safety and efficacy evaluations will be performed as follows:

- Concomitant medications and AEs will be recorded.
- Pain intensity assessed with the Numerical Pain Rating Scale (NPRS), an 11-point scale where 0 is "No Pain" and 10 is "Worst Pain Imaginable: at 0.25, 0.5, 0.75, 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 hours after the administration of study


medication. Assessments between the hours of 00:00 and 06:00 may be skipped if the subject is sleeping; however, consecutive assessments may not be skipped, and the subject must be awakened to complete the Hour 12, Hour 24, and Hour 48 assessments.

- Vital signs: 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 hours after the administration of study medication. Assessments between the hours of 00:00 and 06:00 may be skipped if the subject is sleeping; however, consecutive assessments may not be skipped, and the subject must be awakened to complete the Hour 12, Hour 24, and Hour 48 assessments must be completed even if the subject is asleep.
- Physical exam: 1, 24, and 48 hours after the administration of study medication.
- ECG: 1.5 hours after the administration of study medication.
- Surgical Site assessment: 24 and 48 hours after the administration of study medication.
- Neurosensory Exam of the Foot / Great toe (bilateral): 24 and 48 hours after the administration of study medication.
- Clinical laboratory tests (chemistry/coagulation, hematology, and urinalysis): 1.5 hours after the administration of study medication.
- Blood draw for PK analysis: are at baseline (before dosing), and at 5 minutes, 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, and 48 hours after dosing.

Subjects with inadequately controlled pain may request rescue at any time. However, subjects will be encouraged to receive rescue medication only with an NPRS ≥ 4. Additionally, subjects should be encouraged to wait at least 1 hour after completion of surgery (i.e. completion of sutures) before utilizing pain rescue medication, if possible. Pain intensity (NPRS) will be completed within 15 minutes prior to use of pain rescue medication. While in-clinic, subjects will be treated with the prescribed analgesic regimen (oxycodone 5 mg every 2 hours); however, if subjects do not get adequate analgesic relief they will be discontinued from the efficacy portion of the study. At this point, subjects will receive standard of care analgesics (which may or may not include intravenous opioids). Regardless of discontinuation status, subjects will be followed for safety. Discontinuation affects the computation of the analgesic endpoint only. From Day 3 to 15, over-the-counter standard of care analgesics may be used for management of pain. If needed for management of NPRS score of 4 or higher, oxycodone 5 - 15 mg every 4 - 6 hours.

After completing the assessments through 48 hours after study medication administration, the diary for at-home use will be reviewed and subjects will be discharged from the study center with the diary to record pain assessments and pain medication at home. Subjects will be provided routine standard of care for pain management after discharge from the study center. In their diary, subjects will assess their pain intensity once in the morning (08:00 ±4 hours), and once in the evening (20:00 ±4 hours) using the NPRS. Subjects will also record any medication they take to


treat their pain, and will capture an additional NPRS within 15 minutes prior to each dose of pain medication.

Subjects will return to the study center on Day 8 [±1 day], Day 15 [±2 days] and Day 29 [±2 days], or at the time of discontinuation, for the following assessments: subject home diary review (pain intensity and pain medication at Day 8 and 15 only), in-clinic pain intensity (NPRS), vital signs, surgical site assessment, neurosensory exam of the foot / great toe (bilateral), concomitant medication use, AE assessment, brief pain inventory-short form (BPI-SF), patient global evaluation (PGE), and investigator global evaluation (IGE).

Additionally, on Day 29 [±2 days], or at the time of discontinuation, subjects will have a foot x-ray and a physical exam.

If required due to insufficient wound healing noted at the Day 29 visit, subjects will return to the study center on Day 36 [±2 days] for the following assessments: surgical site assessment, neurosensory exam of the foot / great toe (bilateral), concomitant medication use and AE assessment.

A subject is free to withdraw his/her consent and discontinue participation in the study at any time for any reason.

The protocol-defined visits are presented in Table 2-1:

Table 2-1 Protocol-Specified Visits and Visit Windows

| Study Phase | Visit Time |
|---|---|
| Screening | From days -28 to -1 |
| In-Patient | Days 1 and 2 |
| Follow-up | Days 8(±1 day), 15(±2 days), 29(±2 days) |
| Additional follow-up (if necessary) | Day 36(±2 days) |

#### 2.2.1 Study Population

The study population will consist of 40 healthy subjects between the ages of 18 and 65 years who require bunionectomy.

# 2.2.2 Treatment Regimens

Study Material

The proposed doses of CA-008 to be evaluated in this study are:

- CA-008, 0.5 mg in 10 mL of saline (50 μg/mL)
- CA-008, 1.0 mg in 10 mL of saline (100 μg/mL)
- CA-008, 2.0 mg in 10 mL of saline (200 μg/mL)


- CA-008, 3.0 mg in 10 mL of saline (300 μg/mL)
- CA-008, 4.2 mg in 14 mL of saline (300 μg/mL)

#### **Comparator Group**

• The placebo will be saline for injection.

#### 2.2.3 Treatment Group Assignments or Randomization

The study will be conducted in a double-blinded manner. A computer-generated randomization scheme will be prepared prior to the study start. Subjects who meet the enrollment criteria will be randomly allocated in a 3:1 ratio to receive either active drug or placebo.

Upon enrollment, the site will assign each subject a 3-digit site-specific sequential screening number. The unique subject identification number will consist of a 3-digit original site number followed by a 3-digit screening number. The subject will keep the same number throughout the study. Upon randomization, a unique 4-digit study-specific randomization number will be assigned.

# 2.2.4 Sample Size Determination

The sample size is not based on statistical considerations but is considered appropriate for a Phase 1 dose ranging safety study.

#### 3 GENERAL ANALYSIS AND REPORTING CONVENTIONS

This section discusses general policies to be employed in the analysis and reporting of the data from the study. Departures from these general policies may be provided in the specific detailed sections of this SAP. When this situation occurs, the rules set forth in the specific section take precedence over the general policies.

Each active dose cohort will be presented separately, along with a combined active dose group. Placebo subjects will be pooled across all cohorts in all summaries and analyses.

All continuous study assessments will be summarized by treatment and time point (as applicable) using the descriptive statistics n, mean, SD, median, and range (minimum, and maximum). All of the categorical study assessments will be summarized by treatment and time point (as applicable) using frequency counts and rates of occurrence (%). Changes from baseline for continuous outcomes will be presented as their corresponding continuous measures for post-baseline visits. All study data will be listed by dose cohort, subject, and time point (as applicable).

No preliminary rounding will be performed; rounding will only occur after the analysis. To round, consider the digit to the right of the last significant digit: if <5, then round down; if ≥5, then round up. Means and medians will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one decimal place. A percentage of 100% will be


reported as 100%. Minimums and maximums will be presented with the same precision as the original data.

All analyses will be performed using the SAS System® version 9.3 or higher. The domain (Study data tabulation Model [SDTM]) and analysis (Analysis Data Model [ADaM]) data sets will be taken as input to the SAS programs that generate the report-ready tables, figures and listings. The submission ready SDTM and ADaM data sets will be provided to the sponsor along with display deliveries. The specifications for the domain data sets and analysis data sets will be provided in a separate document.

The following conventions will be used throughout the study analysis:

- Time T0 is the time of completion of study drug administration.
- Assessment visit times are defined by time T0.
- Baseline value is defined as the last valid measurement prior to beginning study drug administration.
- Change from baseline is defined as post-baseline value minus baseline value.
- Duration of an AE will be computed in days for AEs lasting longer than 24 hours, and as hours for AEs lasting less than 24 hours. Duration in hours will be calculated as the stop date/time of the event minus the start date/time. Duration in days will be calculated by using stop date minus the start date +1 if AE occur on or after taking study medication. If AE occur prior to the study medication, then the duration will be calculated by using stop date minus the start date; If reported as ongoing at the time of database lock, the duration will be calculated using the date of the last visit or the last date of any AE for the subject in the database, whichever is later. Missing dates will be imputed as described in Table 8-1.
- The number of days in the study is computed as: [Date of study completion or withdrawal minus the date of study drug administration (Day 1)] + 1.
- If duplicate values are obtained at a given visit (e.g., repeated vital sign
  measurements), the last value will be used unless it is noted that the measurement
  was in error for that value. Values that compromise interpretation will not be used in
  summaries (e.g., values that were obtained post-dose will not be summarized as predose values).
- If a pre-rescue NPRS is recorded in the same minute as a rescue medication is recorded, the NPRS will be assumed to have occurred PRIOR to the administration of rescue.
- If a subject experiences inadequate analgesic relief and are discontinued from the efficacy portion of the study the date/time of the discontinuation will be assumed to be the date/time of the start of standard of care analgesic rescue.

#### 4 SUBJECT POPULATIONS

#### 4.1 Analysis Populations


Two analysis populations are defined as follows:

 Safety Population will include all randomized subjects who received any amount of study drug

 Pharmacokinetic (PK) population: All randomized participants who received any amount of study drug and have sufficient plasma concentrations for estimation of at least one PK parameter.

Membership in the safety analysis population will be determined before unblinding any study treatment codes. Membership in the PK analysis population will be determined after unblinding and receipt of the PK concentration and PK parameter data from the analytical lab. For all analyses, subjects will be analyzed by treatment group according to the actual product received during treatment, i.e., "as treated."

# 4.2 Disposition of Subjects

All subjects and the populations for which they qualify will be listed. Subjects who are screened and who fail screening or withdraw consent prior to randomization or are randomized but not treated will be listed and summarized in the disposition summary table. Subjects who are randomized, subject inclusion into each study population, subjects who are treated, subjects who complete follow-up as well as subjects who withdraw early from the study and the reason for withdrawal will be summarized by treatment group and overall in the subject disposition summary table. Subjects who are discontinued from the efficacy portion of the study will also be presented.

A listing of CRF comments by time point and CRF section will also be presented.

#### 4.3 Protocol Deviations

Deviations are categorized as informed consent procedures, inclusion/exclusion criteria, study medication, prohibited medications, study procedures, study drug assignment/treatment, visit or assessment time window, missed visit or assessment and/or other. All protocol deviations will be captured on CRFs and documented in site specific logs throughout the study. Deviations will be categorized and classified as major or minor by the project team and the medical monitor after database lock but before unbinding, and will be discussed in the CSR. The number of subjects with protocol deviations, both minor and major, will be presented in a data listing and will be summarized by type of deviation and major/minor classification.

#### 5 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

#### 5.1 Demographics and Baseline Characteristics

Demographic variables include age, sex, race, and ethnicity. Baseline characteristics include American Society of Anesthesiologists (ASA) physical status, height, weight (kg), and BMI (kg/m²). Demographics and baseline characteristics will be presented in a by-subject listing and summarized overall and by treatment group.


#### 5.2 Medical/Surgical History

Medical and Surgical history, as collected at screening, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 20.1 to determine system organ class (SOC) and preferred term (PT). Medical histories will be presented in a by-subject listing.

Any events that occur prior to the study procedure will be categorized as medical history.

#### **5.3** Prior and Concomitant Medications

Prior medications/therapies are those that stop prior to the start of the study drug administration. Any medication/therapy that stops at or after this time or with missing stop dates is considered concomitant medication/therapy.

Prior and concomitant medications are collected at screening and updated throughout the study as needed. Prior and concomitant medications will be coded using WHO/ATC classification index version September 2017. The number and percentage of subjects who take concomitant medications will be summarized by drug class and preferred term, overall and by treatment group, for the safety population.

All medications and non-medical therapies captured in CRFs will appear in data listings.

#### 6 MEASUREMENTS OF TREATMENT EXPOSURE and COMPLIANCE

Because study medication is administered as a single dose at the study center by trained study personnel, compliance with respect to study medication will not be calculated. A listing of study drug administration and exposure data will be provided.

After completing the assessments through 48 hours after study medication administration, the diary for at-home use will be distributed to the subject to collect pain intensity (twice daily on NPRS) and pain medication through Day 15. Compliance with home diary use will be evaluated based on post-discharge home diary records. Compliance for each subject will be based on the number of days the subject participated in the outpatient study period, defined as:

Where the N of expected NPRS records in the diary for each subject is calculated as 2 times the number of days the subject participated in the outpatient portion of the study. The number of days of participation will be calculated as the date of the Day 15 visit or the date of the last study visit (whichever is earlier) minus the date of discharge. NPRS recorded prior to a rescue use will not be included in this calculation of compliance.

For example, Subject A was discharged on Day 2, if this subject discontinues the study on Day 18, then the expected N of NPRS records on diary will be 36 (2 \* (15-2)). Assuming Subject A had CONFIDENTIAL


Sponsor: Concentric Analgesics, Inc.

Statistical Analysis Plan Protocol Number: CA-PS-2017-101 Date: 31Mar2018

10 NPRS available from his/her diary, then compliance for this subject would be 27.8% ((10/36) \*100). However, if subject A had discontinued the study on Day 10 (prior to Day 15), then the expected N of NPRS for this subject would be 16 (2 \* (10-2)) and compliance would be 62.5 % ((10/16) \*100). A summary of compliance will be provided overall and by treatment group.

Compliance with recording an NPRS prior to rescue in the diary will be calculated as the number of NPRS recorded prior to taking rescue medications divided by the number of rescue medication uses recorded.


#### 7 EFFICACY EVALUATION

# 7.1 Handling of Dropouts or Missing Data

All efforts will be made to minimize missing data. These efforts will include the following:

- Subjects are required to consent to continuous data collection even after discontinuation of study medication;
- Data collection will continue after subjects take rescue medication.

With the procedures above, it is expected that missing data will be minimal. Missing at random is expected to be a reasonable assumption for this dose-escalation study.

For subjects who take protocol allowed rescue medication a windowed last pain score carried forward (LOCF) will be used. The pre-rescue pain score will be used to impute scheduled assessments for 4 hours following the rescue use. Intermittent missing pain scores (due to subject sleeping, etc.) will not be imputed, and AUC will be calculated based on non-missing values. For subjects who drop out of the study prior to Day 15, or who are discontinued from efficacy and given SOC analgesics for inadequate pain relief, scheduled assessments will first be imputed using the worst prior pain score carried forward (WOCF) using the worst scheduled non missing pain score prior to drop out within the AUC period being calculated (e.g., if the AUC being calculated includes hours 12-24, the worst observed pain score between hours 12 and 24 will be used). As a sensitivity, the AUC will also be calculated where assessments after drop out will be imputed using LOCF, using the last scheduled non missing pain score prior to drop out.

#### 7.2 Assessment Time Windows

Safety assessment summaries will be based on the nominal protocol-specified assessment times. NPRS scores will be based on actual collection dates/times wherever possible. If no collection date/time is available the nearest protocol specified assessment time will be used.

## 7.3 Exploratory Efficacy Endpoints

- Area under the curve (AUC) of subject's NPRS will be examined over various time periods, including but not limited to: AUC(0-12), AUC(12-24), AUC(24-48), AUC(24-72), AUC(24-96), AUC(24h to Week 1), and AUC(24h to Week 2).
- Mean daily opioid consumption (in morphine equivalents) over the same time periods as the AUC calculations above.
- Proportion of patients who drop out of the study due to inadequate analgesia from Day 1 to 15.
- Brief Pain Inventory-short form (BPI-SF) scores at the Day 8 (Week 1), Day 15 (Week
   2) and Day 29 (Week 4) or ET clinic visits.
- Patient Global Evaluation (PGE) at the Day 8 (Week 1), Day 15 (Week 2) and Day 29 (Week 4) clinic visits.


Sponsor: Concentric Analgesics, Inc.

Protocol Number: CA-PS-2017-101

Date: 31Mar2018

 Investigator Global Evaluation (IGE) at the Day 8 (Week 1), Day 15 (Week 2) and Day 29 (Week 4) clinic visits.

- Time to first use of rescue medication.
- Percent of days that rescue medication was used.

# 7.4 Analysis Methods

Formal hypotheses testing will be not conducted. All p-values will be considered nominal in this study and no adjustments for multiplicity will be performed. All efficacy analyses will be based on the safety population.

#### 7.4.1 AUC Outcomes

All AUC calculations will be done using the standard trapezoidal rule

AUC = 
$$\sum_{i=0}^{x} \left( \frac{NPRS_i + NPRS_{i+1}}{2} \right) * (T_{i+1} - T_i)$$

Where: NPRS<sub>i</sub> = NPRS at time i, and  $(T_{i+1} - T_i)$  is the Time difference in hours between time i and time i+1.

Missing NPRS will be handled as discussed in Section 7.1.

AUC values will be analyzed using a 1-factor (treatment) analysis of variance (ANOVA) model with treatment as the main effect. In addition to the individual comparisons between each of the five CA-008 groups and the placebo group, the test for a linear trend across dose groups will be carried out using the scores 0, 0.5, 1.0, 2.0, 3.0 and 4.2 for the placebo group and the five active groups, respectively.

The AUC analyses will be presented in a summary table with standard summary statistics for each dose cohort and placebo as well as active vs. placebo mean differences, standard errors, confidence intervals and comparison p-values as appropriate. Comparisons of individual dose cohorts for dose response may be presented for certain secondary AUC endpoints.

Mean NPRS scores over time (in-clinic and diary) will be graphed over time by dose cohort. NPRS over time by each subject may also be displayed graphically as warranted. The individual NPRS and the computed AUC variables will be listed for all individual subjects.

#### 7.4.2 Average Daily NPRS score of 2 daily diary assessments

The Average Daily NPRS scores will be computed for each subject using the NPRS scores recorded in the take-home diary from study days 3-15.

The Average Daily NPRS will be the average of the AM and PM scores within each day. If individual AM or PM NPRS scores are missing, the score that is present will be used as the daily average. If both scores are missing for any day, then that day will not have a daily average. The mean across all subjects of the average daily scores on each day will be graphed by day and


dose cohort. If rescue medication was taken within 4 hours of the AM or PM PI assessment, it will be replaced with the pre-rescue NPRS (if available) in the daily average.

The average daily NPRS scores will be analyzed using the same type of ANOVA model as described in Section 7.4.1 at each time point. In addition, actual date/time NPRS assessed over the outpatient period from T48h onward will be used to calculate AUC between 24 hours and Week 1 and between 24 and Week 2 and compared versus placebo.

#### 7.4.3 Total daily opioid consumption (in oral morphine equivalents)

The amount of opioids taken as rescue will be calculated using the rescue medication page of the eCRF. If additional opioids, other than the study rescue medications, appear on the concomitant medications page and can be identified, those opioids will also be included (in terms of morphine equivalents) in the total consumed. For summaries of opioid consumption, the rescue medications for subjects who are discontinued from the efficacy portion of the study will be counted two ways. First, all medications on days up to and including the date of the discontinuation from efficacy will be included, but medications that were continued after the date of discontinuation from efficacy will not be counted. In a second analysis, all the medication for these subjects will be counted, regardless of whether it was taken before or after the subject discontinued from the efficacy portion.

Table 7-1 will be used to calculate the morphine milligram equivalents (MEQ) for each medication. The total opioid consumption for each day for each subject will be calculated as the sum of the MEQs of all of the medications taken on that day. For example, if a subject takes 5 MEQ morphine on Day 1 and Day 2, and 10 MEQ of Oxycodone on Day 2, the total consumption for Day 1 is 5 MEQ, and the total consumption for Day 2 is 15 MEQ. Subjects that take no opioids on a day will have a total opioid consumption value of zero for that day.

Table 7-1 Table of Morphine Milligram Equivalents

(from cdc.gov/drugoverdose/pdf)

| Opioid (Doses in mg/day) | Conversion Factor |
|----------------------------------|-------------------|
| Codeine | 0.15 |
| Fentanyl transdermal (in mcg/hr) | 2.4 |
| Hydrocodone | 1 |
| Hydromorphone | 4 |
| Morphine | 1 |
| Oxycodone | 1.5 |
| Oxymorphone | 3 |


Total opioid consumption will be calculated overall and for the same periods as the NPRS AUC values: 0-12 hours, 12-24 hours, 24-48 hours, 24-72 hours and 24-96 hours in addition, the periods 24h to Week 1 and 24h to Week 2 will also be summarized. An ANOVA with treatment arm as the main effect will be performed and the same types of comparisons as described in Section 7.4.1 will be presented. A separate summary containing only subjects that have taken at least one dose of rescue will be performed if warranted.

# 7.4.4 Proportion of patients who drop out of the study due to inadequate analgesia from Day 1 to 15.

Proportion of subjects who drop out of the study due to inadequate analgesia from Day 1 to 15 will be analyzed using Fisher's exact tests. Inadequate analgesia will be assumed if a subject drops out of the efficacy portion of the study due to inadequate analgesia, or if a subject drops out of the study entirely due to lack of efficacy or for an AE that is pain related. The reasons for discontinuation as documented on the eCRF end of study page will be used to determine the subjects who drop out of the study for inadequate analgesia.

A summary table will present the active vs. placebo group proportions, 95% confidence intervals and two-sided Fisher's exact p-values for the difference in proportions between each active group and placebo.

### 7.4.5 Brief Pain Inventory-short form (BPI-SF)

Individual questions will be listed.

In addition, two sub scores of the BPI will be calculated as follows:

Pain Severity Score = Mean of items 3-6

Pain Interference Score = Mean of items 9A-9G calculated only if more than 50%, or four of seven, of the total items have been completed on a given administration.

Questions 3-6, the Pain Severity Score and the Pain Interference Score will be analyzed using ANOVA with treatment as the main effect similar to previous analyses. The analysis results will be presented in a summary table with active vs. placebo difference means, standard errors, confidence intervals and p-values.

#### 7.4.6 PGE and IGE

The proportions of subjects in each individual PGE and IGE category will be summarized by treatment group and time point and analyzed using the Cochran-Mantel-Haenszel mean score test (using equally spaced scores) at each time point to compare treatments across the 4 levels of outcomes (poor, fair, good, or excellent). In addition, Fisher's exact test will be performed to compare treatments across 2 levels of outcomes (Poor/Fair versus Good/excellent). The continuous PGE and IGE scores will also be analyzed using ANOVA with treatment as a main effect similar to presented previously. Individual PGE and IGE scores will be listed.


#### 7.4.7 Time to First Use of Rescue Medication

The time to first rescue will be measured from Time 0 (time of completion of study drug administration). If a subject does not take rescue medication but prematurely discontinues from the study or discontinues from the efficacy portion of the study, then for analysis purposes the subject's observation time will be the time of the discontinuation. For subjects who discontinue from the efficacy portion of the study, the discontinuation time will be considered to be a rescue event. The time will be considered to be a rescue event if the discontinuation from the study was due to lack of efficacy, otherwise, it will be considered a censored observation.

The distributions of time to first rescue in each treatment group will be presented graphically using Kaplan-Meier plots.

If data warrant, a summary table will present the number of subjects receiving rescue medication, number of censored subjects, median time to first dose of rescue, and 95% confidence intervals of the medians by dose cohort. Individual times to event will be listed.

#### 7.4.8 Percent of Subjects Taking Rescue / Use of Rescue Medication over Time

Subjects will be counted as having taken rescue on any particular day based on the rescue medication page of the eCRF and the at home rescue diary. If additional medications, other than the study rescue medications, appear on the concomitant medications page and can be identified as having been taken for bunion pain, those medications will also be counted.

The proportion of subjects taking rescue will be summarized for each study day through Day 15. For summaries, subjects who discontinued from the efficacy portion of the study will be counted two ways. First, all medications on days up to and including the date of the discontinuation from efficacy will be included, but medications that were continued after the date of discontinuation from efficacy will not be counted. In a second analysis, all the medication for these subjects will be counted, regardless of whether it was taken before or after the subject discontinued from the efficacy portion.

In addition, the proportion of subjects taking any rescue medication during the following periods: 0 to 48 hours, 0 to 72 hours, 0 to 96 hours, Days 1 to 8, Days 3-8, and Days 9-15 and overall will be summarized and will be analyzed using Fisher's exact tests.

Separate summaries for opioid and non-opioid rescue use will be presented if sufficient data are present in the groups.

#### **8 SAFETY EVALUATION**

#### 8.1 Overview of Safety Analysis Methods

All safety outcomes will be summarized using the safety population. Safety outcomes include:

- Incidence of TEAEs
- Clinical laboratory test results


- Vital sign measurements
- Electrocardiogram (ECG) results
- Physical Exam findings
- Surgical Site assessment findings
- Neurosensory Exam results

#### 8.2 Adverse Events

Any untoward medical event that occurs after signing the ICF is considered to be an adverse event (AE). Treatment-emergent AEs are defined as AEs that start or worsen in severity after the first exposure to study drug and up to Day 29 for non-SAEs (up to Day 59 for SAEs). Verbatim terms used by investigators to identify AEs in the CRFs will be mapped to the appropriate preferred term (PT) and system organ class (SOC) using a standardized coding dictionary (MedDRA Version 19.1). All coding will be reviewed prior to database lock. All recorded AEs will be listed, but only TEAEs will be summarized.

For evaluation of causal relatedness to treatment, the categories are probably related, possibly related or unlikely related. For categorization in the summary tables, AEs designated as probably or possibly related will be considered to be related.

For the evaluation of event severity terms, the criteria are mild, moderate, severe or life-threatening.

In addition to a listing of all TEAEs, treatment related TEAEs, serious TEAEs, Deaths, and TEAEs leading to premature discontinuation from the study will be provided.

An overall summary will be prepared giving for each treatment group and overall both the number of TEAEs, and the number of subjects with TEAEs, as well as SAEs, treatment related TEAEs and TEAEs leading to premature discontinuation from study.

The number of subjects with AEs will be summarized for each treatment group by SOC and PT sorted in alphabetically by system organ class (SOC), and then by preferred term (PT) within SOC. These summaries will be given by treatment in separate tables for each of the following TEAE event sets:

- All events
- Treatment related events
- Serious events
- Events leading to premature discontinuation from study
- Events by maximum severity

If a given subject experiences a TEAE that maps to the same PT/SOC more than once, the subject will be counted only once for the SOC/PT at the greatest severity (i.e., mild, moderate, or severe) and causality (i.e., attribution to study material).


Duration of a TEAE lasting more than 24 hours will be computed in days as the stop date of the event minus the start date plus 1 and will be reported in days. TEAEs lasting less than 24 hours will be computed as stop date/time minus start date/time. If reported as ongoing at the time of database lock, the stop date is defined as the date of the last visit or the last date of any event for the subject in the database, whichever is later. If a TEAE is considered resolved, but the stop date is missing, the last day of the month will be imputed if the month and year are available. If only the year is available, and the year is the same as the year of the last visit, the stop date will be the latest of the last visit date or latest event for the subject in the database. If the year of the event is prior to the year of the last treatment, the end day and month will be set to 31 December.

For missing or partial start and stop dates/times, the most conservative imputation will be used (AEs will be assumed to be temporally related to the study medication). Table 8-1 will be used to impute any missing dates/times:

Table 8-1 Table of Imputation Rules for Missing AE Start Dates

| Missing Date<br>Portion | Prior to<br>Treatment | Same as Treatment<br>Start Date | After Treatment Start<br>Date |
|---|---|---|---|
| Day | Month and Year <<br>Month and Year of<br>Study treatment: | Month and Year =<br>Month and Year of<br>Study treatment: | Month and Year ><br>Month and Year of<br>Study Treatment: |
| | Start Day = 1 Stop Day=last day of | Start Day = Day of first<br>treatment | Start Day = 1<br>Stop Day=last day of |
| | the month | Stop Day= last day of the month | the month |
| Day and Month Define Day as | Year < Year of first treatment: | Year = Year of study<br>treatment: | Year > Year of study<br>treatment: |
| above, then: | Start Month = July | Start Month = Month of<br>study treatment | Start Month = January |
| | Stop Month = Dec | Stop Month = Dec | Stop Month = Dec |
| Day, Month, and<br>Year | 1 | | |
| Time Missing start times will be imputed as 00:01 | | e imputed as 00:01 | |
| Missing stop times will be imputed as 11:59 | | | |

After following these imputation rules, if the start date/time is imputed as a date after the end date/time, the start date/time will be set to the end date/time to provide a positive duration for the event incidence.


Missing assessments for AE study medication relationship or severity will be analyzed as related or severe respectively. No other imputation is planned for safety data.

## 8.3 Clinical Laboratory Evaluation

Clinical laboratory test results (blood chemistry/coagulation, hematology and urinalysis) will be listed for individual subjects. Baseline for clinical laboratory parameters will be defined as the last evaluation before dosing with study treatment. For each individual lab test value, the raw value and change from baseline will be summarized by treatment and time point.

Each clinical laboratory test will be defined by the clinical laboratory to be "Low", "Normal", or "High", according to the normal reference range from the clinical laboratory. The number and percentage of subjects who have a shift from within to outside the normal reference range from baseline (and vice versa) to each follow-up visit will be summarized by treatment and time point.

## 8.4 Vital Signs

Vital signs results including BP (systolic and diastolic), pulse rate, respiration rate, and body temperature will be listed for individual subjects. Baseline for vital signs measurements will be defined as the last evaluation before dosing with study medication. Summary statistics, including change from baseline, will be determined for each measure and will be summarized by treatment and time point.

#### 8.5 Physical Examination

Physical examination abnormality results will be listed for individual subjects.

#### 8.6 Surgical Site Assessment

The surgical site abnormality results and assessment score results will be listed and will be summarized by treatment and visit.

# 8.7 Neurosensory Assessment

The neurosensory assessment results will be listed and the number of subjects with normal/abnormal assessments will be summarized descriptively by treatment and time point.

#### 8.8 ECG Examinations

ECG examination abnormality results will be listed for individual subjects and number of subjects with abnormal results will be summarized descriptively by treatment and time point.

#### 8.9 Drugs of Abuse and Alcohol Screens, Pregnancy Test.


Pregnancy (for female subjects of childbearing potential), urine drug screen and alcohol breath tests will be performed at screening and pre-procedure. Results will be listed for individual subjects. Each test result will be defined to be "negative" or "positive".

## 8.10 Patient Pain Assessment Training and Surgery Details

Patient pain assessment training and surgery details will be documented in CRFs and will be listed for each subject.

#### 9 PHARMACOKINETIC EVALUATION

Blood draws for PK analysis will be done at baseline (before dosing), and at 5 minutes, 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, and 48 hours after dosing. Blood levels of CA-008, CA-101, capsaicin and capsaicin glucuronide metabolite will be determined. PK sample collections and drug levels will be listed.

There will be a separate PK Analysis Plan that will describe the analyses of all PK concentrations.


#### 10 OTHER ANALYSES

Any additional analyses not included in this SAP conducted after database lock will be considered exploratory and identified as Post Hoc in the CSR.

#### 11 INTERIM ANALYSES AND DATA MONITORING

There are no planned interim analyses for this study.

A DMC will regularly monitor safety data in a blinded fashion throughout the study. To determine appropriate dose escalation in the next planned cohort, safety data will be reviewed by a DMC after the final dosing within each cohort. Details regarding the DMC are included in the DMC Charter.

#### 12 CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL

Any deviations from the statistical plan will be described and a justification given in the CSR.

#### 13 REFERENCES

US Federal Register. (1998) International Conference on Harmonization; Guidance for Industry: Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration. Federal Register, Vol. 63, No. 179, September 16, 1998, page 49583.

US Federal Register. (1996) International Conference on Harmonization; Guidance for Industry: Structure and Content of Clinical Study Reports. Department of Health and Human Services: Food and Drug Administration. Federal Register Vol. 61, July 17, 1996, page 37320.

Guidance for Industry (2014) Analgesic Indications: Developing Drug and Biological Products - Draft Guidance. Department of Health and Human Services: Food and Drug Administration. Center for Drug Evaluation and Research (CDER) February 2014 Clinical/Medical.


# 14 APPENDICES

# 14.1 Tables, Figures and Listings for Final Study Report

# 14.1.1 Tables

| Table 14.1.1 | All Subjects | Summary of Subject Disposition |
|---|---|---|
| Table 14.1.2 | All Randomized Population | Summary of Protocol Deviations |
| Table 14.1.3 | All Randomized Population | Summary of Demographic and Baseline Characteristics |
| Table 14.1.4 | Safety Population | Summary of Concomitant Medications by ATC Class and Preferred Term |
| Table 14.1.5 | Safety Population | Summary of Subject NPRS and NPRS at Rescue Diary Compliance |
| Table 14.2.1.1 | Safety Population | ANOVA Analysis of AUC of NPRS - WOCF |
| Table 14.2.1.2 | Safety Population | ANOVA Analysis of AUC of NPRS - LOCF |
| Table 14.2.2.1 | Safety Population | ANOVA Analysis Mean Average Daily NPRS of 2 Daily Diary Assessments |
| Table 14.2.3.1.1 | Safety Population | Summary of Daily Opioid Consumption (in Morphine equivalents) by Study Day |
| Table 14.2.3.1.2 | Safety Population | Summary of Daily Opioid Consumption (in Morphine equivalents) by Study Day up to Discontinuation of Efficacy Portion |
| Table 14.2.3.2.1 | Safety Population | ANOVA Analysis Mean Daily Opioid Consumption (in Morphine Equivalents) |
| Table 14.2.3.2.2 | Safety Population | ANOVA Analysis Mean Daily Opioid Consumption (in Morphine Equivalents) up to Discontinuation of Efficacy Portion |
| Table 14.2.3.3 | Safety Population –<br>Subjects Who Took<br>Any Opioid<br>Medication | ANOVA Analysis Mean Daily Opioid Consumption (in Morphine Equivalents) |
| Table 14.2.4 | Safety Population | Fishers Analysis of Proportion of Drop Out Due to Inadequate Analgesia |
| Table 14.2.5 | Safety Population | ANOVA Analysis Brief Pain Inventory (BPI-SF) Pain and Interference Subscales |


| Table 14.2.6 | Safety Population | CMH and Fishers Analysis of Patient Global Evaluation (PGE) |
|---|---|---|
| Table 14.2.7 | Safety Population | CMH and Fishers Analysis of Investigator Global Evaluation (IGE) |
| Table 14.2.8.1.1 | Safety Population | Fishers Analysis of Percent of Subjects using Rescue Medication Over Time |
| Table 14.2.8.1.2 | Safety Population | Fishers Analysis of Percent of Subjects using Rescue<br>Medication Over Time up to Discontinuation of Efficacy<br>Portion |
| Table 14.2.8.2.1 | Safety Population | Summary of Percent of Subjects Using Rescue<br>Medication by Day |
| Table 14.2.8.2.2 | Safety Population | Summary of Percent of Subjects Using Rescue<br>Medication by Day up to Discontinuation of Efficacy<br>Portion |
| Table 14.2.9 | Safety Population | Kaplan-Meier Analysis of Time to First Use of Rescue Medication by Dose (if needed) |
| Table 14.3.1.1 | Safety Population | Overall Summary of Treatment-Emergent Adverse Events (TEAEs) |
| Table 14.3.1.2 | Safety Population | Summary of TEAEs by System Organ Class and Preferred Term |
| Table 14.3.1.3 | Safety Population | Summary of Treatment Related TEAEs by System Organ Class and Preferred Term |
| Table 14.3.1.4 | Safety Population | Summary of SAEs by System Organ Class and Preferred Term |
| Table 14.3.1.5 | Safety Population | Summary of TEAEs Leading to Discontinuation from Study |
| Table 14.3.1.6 | Safety Population | Summary of TEAEs by System Organ Class, Preferred Term and Severity |
| Table 14.3.1.7 | Safety Population | Summary of TEAEs by System Organ Class, Preferred Term and Relationship to Study Drug |
| Table 14.3.2.1.1 | Safety Population | Summary of Blood Chemistry/Coagulation Laboratory<br>Tests: Results and Change from Baseline |
| Table 14.3.2.1.2 | Safety Population | Summary of Blood Chemistry/Coagulation Laboratory<br>Tests: Shifts from Baseline |
| Table 14.3.2.2.1 | Safety Population | Summary of Hematology Laboratory Tests: Results and Change from Baseline |
| Table 14.3.2.2.2 | Safety Population | Summary of Hematology Laboratory Tests: Shifts from Baseline |
| Table 14.3.2.3.1 | Safety Population | Summary of Urinalysis Laboratory Tests: Results and Change from Baseline |


| Table 14.3.2.3.2 | Safety Population | Summary of Urinalysis Laboratory Tests: Shifts from Baseline |
|---|---|---|
| Table 14.3.4 | Safety Population | Summary of Vital Signs: Results and Change from Baseline |
| Table 14.3.5 | Safety Population | Summary of Surgical Site Assessment |
| Table 14.3.6.1 | Safety Population | Summary of Neurosensory Exam –Target Foot |
| Table 14.3.6.2 | Safety Population | Summary of Neurosensory Exam –Non-Target Foot |
| Table 14.3.7 | Safety Population | Summary of ECG Exam Abnormal Findings |

# 14.1.2 Figures

| Figure 14.2.1.1 | Safety Population | Mean NPRS Over Time by Treatment (WOCF) |
|---|---|---|
| Figure 14.2.1.2 | Safety Population | Mean NPRS Over Time by Treatment (LOCF) |
| Figure 14.2.2 | Safety Population | Mean NPRS Over Time by Subject (Observed Data, no imputation for Drop Out) |
| Figure 14.2.3 | Safety Population | Average Daily NPRS of 2 Daily Diary Assessments by Treatment |
| Figure 14.2.4 | Safety Population | Time to First Use of Rescue Medication |

# 14.1.3 Listings

| Listing 16.2.1 | All Subjects | Informed Consent, Randomization and Study Population |
|---|---|---|
| Listing 16.2.2 | All Randomized<br>Subjects | Eligibility |
| Listing 16.2.3 | All Randomized<br>Subjects | Protocol Deviations |
| Listing 16.2.4 | All Randomized<br>Subjects | Subject Completion/Early Termination |
| Listing 16.2.5 | All Randomized<br>Subjects | Demographics and Baseline Characteristics |
| Listing 16.2.6 | All Randomized<br>Subjects | Medical/Surgical History |
| Listing 16.2.7.1 | All Randomized<br>Subjects | Prior and Concomitant Medications |
| Listing 16.2.7.2 | All Randomized<br>Subjects | Rescue Medication Administration |
| Listing 16.2.7.3 | All Randomized<br>Subjects | Non-Medication Therapies |


| Listing 16.2.7.4 | All Randomized<br>Subjects | Time to First Use of Rescue Medication and AUC of Total MEQ |
|---|---|---|
| Listing 16.2.8 | All Randomized<br>Subjects | X-Ray of Surgical Site |
| Listing 16.2.9 | All Randomized<br>Subjects | Bunionectomy Surgery |
| Listing 16.2.10 | All Randomized<br>Subjects | Study Drug Administration |
| Listing 16.2.11 | All Randomized<br>Subjects | Subject NPRS and NPRS at Rescue Diary Compliance |
| Listing 16.2.12 | All Randomized<br>Subjects | Discharge from Clinic |
| Listing 16.2.13 | All Randomized<br>Subjects | Paper Diary Collection |
| Listing 16.2.14.1 | All Randomized<br>Subjects | Pain Intensity Assessment (NPRS) |
| Listing 16.2.14.2 | All Randomized<br>Subjects | AUC of Pain Intensity Assessment (NPRS) - WOCF |
| Listing 16.2.14.3 | All Randomized<br>Subjects | AUC of Pain Intensity Assessment (NPRS) - LOCF |
| Listing 16.2.15.1 | All Randomized<br>Subjects | Brief Pain Inventory (BPI-SF) – Pain Scale |
| Listing 16.2.15.2 | All Randomized<br>Subjects | Brief Pain Inventory (BPI-SF) – Pain Interference |
| Listing 16.2.16 | All Randomized<br>Subjects | Patient Global Evaluation (PGE) |
| Listing 16.2.17 | All Randomized<br>Subjects | Investigator Global Evaluation (IGE) |
| Listing 16.2.18.1 | All Randomized<br>Subjects | Adverse Events |
| Listing 16.2.18.2 | All Randomized<br>Subjects | Serious Adverse Events |
| Listing 16.2.18.3 | All Randomized<br>Subjects | Treatment Related Adverse Events |
| Listing 16.2.18.4 | All Randomized<br>Subjects | Adverse Events Leading to Premature Study Discontinuation |
| Listing 16.2.19.1 | All Randomized<br>Subjects | Blood Chemistry/Coagulation Laboratory Results |
| Listing 16.2.19.2 | All Randomized<br>Subjects | Hematology Laboratory Results |


| Listing 16.2.19.3 | All Randomized<br>Subjects | Urinalysis Laboratory Test Results |
|---|---|---|
| Listing 16.2.20 | All Randomized<br>Subjects | Alcohol Breath and Urine Drug Screen Tests |
| Listing 16.2.21 | All Randomized<br>Subjects | Pregnancy Test |
| Listing 16.2.22 | All Randomized<br>Subjects | Vital Signs |
| Listing 16.2.23 | All Randomized<br>Subjects | Physical Exam and Brief Physical Exam Assessment |
| Listing 16.2.24 | All Randomized<br>Subjects | Surgical Site Assessment |
| Listing 16.2.25 | All Randomized<br>Subjects | Neurosensory Exam |
| Listing 16.2.26 | All Randomized<br>Subjects | 12-Lead Electrocardiogram |
| Listing 16.2.27 | PK Population | Pharmacokinetic (PK) Concentration Data |




# **Certificate Of Completion**

Envelope Id: 425E9A5818E343B58B90E816481BA9E7

Subject: Please DocuSign: CA-PS-2017-101 SAP Final v2.0 31Mar2018.pdf

Source Envelope:

Document Pages: 32 Signatures: 3 Envelope Originator: Certificate Pages: 4 Initials: 0

AutoNav: Enabled

Envelopeld Stamping: Enabled

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

Caitlyn Avila

Pasadena, CA 91105

Status: Completed

100 W California Blvd., Unit 25

cavila@lotuscr.com IP Address: 205.197.253.4

# **Record Tracking**

Status: Original

4/2/2018 9:19:48 AM

Holder: Caitlyn Avila cavila@lotuscr.com Location: DocuSign

#### Signer Events

Jennifer Nezzer inezzer@lotuscr.com **Director of Biometrics** 

Lotus Clinical Research

Security Level: Email, Account Authentication

(Required)

#### Signature

Jennifer Neyyer

**Timestamp** 

Sent: 4/2/2018 9:21:17 AM Viewed: 4/2/2018 7:09:58 PM Signed: 4/2/2018 7:10:20 PM

Signature ID:

F51546CD-923C-410C-87CA-B1F62D450C79

Using IP Address: 45.18.125.80

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I have reviewed this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 8/16/2017 8:46:58 AM

ID: a2e3d9e3-0ef1-4b5e-8f0a-26d3d9799cc6

Pob Allen

Sent: 4/2/2018 9:21:17 AM Resent: 4/5/2018 9:33:40 AM Viewed: 4/5/2018 4:15:37 PM Signed: 4/5/2018 4:16:31 PM

Rob Allen

rob@concentricanalgesics.com

Concentric Analgesics

Security Level: Email, Account Authentication

(Required)

Signature ID:

EF39BEAA-FE45-423B-BCF8-D0AF4EA284B3

Using IP Address: 71.230.253.85

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 10/13/2017 11:50:20 AM

ID: 2878f2a9-ac54-4c02-a6e2-cc535239d936

Song lion

Sent: 4/2/2018 9:21:16 AM Viewed: 4/2/2018 9:23:25 AM Signed: 4/2/2018 9:24:09 AM

Song Liou

sliou@lotuscr.com

Lotus Clinical Research

Security Level: Email, Account Authentication (Required)

Signature ID:

85C80776-CFA1-404F-B9C3-4B43BB0AA100

Using IP Address: 108.51.237.84

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I am the author of this document

**Electronic Record and Signature Disclosure:** 

| Accepted: 2/16/2018 10:40:34 AM | • | • |
|---|---|---|
| ID: 33003533-520a-46d0-b1ac-311cccf15c53 | | |
| In Person Signer Events | Signature | Timestamp |
| | o.ga.a. | <b>p</b> |
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| | | • |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| , | | |
| Carbon Copy Events | Status | Timestamp |
| Notary Events | Signature | Timestamp |
| | | , <b>,</b> |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 4/5/2018 9:33:40 AM |
| Certified Delivered | Security Checked | 4/5/2018 4:15:37 PM |
| Signing Complete | Security Checked | 4/5/2018 4:16:31 PM |
| Completed | Security Checked | 4/5/2018 4:16:31 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

Timestamp

Signature

Signer Events

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

Please read the information below carefully and thoroughly. By checking the "I agree to use Electronic Records and Signatures" box in the DocuSign system, you confirm you can access this information electronically to your satisfaction and agree to these terms and conditions below.

# **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after signing session. If you wish for us to send you paper copies of any such documents from our office to you, please contact your Lotus Lead Project Manager.

# Withdrawing your consent

If you decide to receive documents from us electronically, you may at any time change your mind and tell us thereafter that you want to receive documents only in paper format. If you want to withdraw your consent and receive future documents in paper format, please contact your Lotus Lead Project Manager.

# Consequences of changing your mind

If you elect to receive documents only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the documents to you in paper format, and then wait until we receive back from you and your execution of such paper documents. To indicate to us that you are changing your mind within the DocuSign system, you must withdraw your consent using the DocuSign "Withdraw Consent" form on the signing page of a DocuSign envelope instead of signing it. This will indicate to us that you have withdrawn your consent to receive documents electronically from us and you will no longer be able to use the DocuSign system to receive documents electronically from us or to sign electronically documents from us.

# All documents will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all documents that require your signature during the course of our relationship with you. All documents will be sent to you through your e-mail as recorded in the study-specific Study Contact Sheet. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# How to contact Lotus Clinical Research, LLC:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically:

#### To advise Lotus Clinical Research, LLC of your new e-mail address

To let us know of a change in your e-mail address, you must send an email message to your Lotus Lead Project Manager and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.

In addition, you must notify DocuSign, Inc. to arrange for your new email address to be reflected

in your DocuSign account by following the process for changing e-mail in the DocuSign system.

# To request paper copies from Lotus Clinical Research, LLC

To request delivery from us of paper copies of the documents previously provided by us to you electronically, you must send an e-mail to your Lotus Lead Project Manager and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number.

## To withdraw your consent

To inform us that you no longer want to receive future documents in electronic format via DocuSign you may:

i. decline to sign a document from within your DocuSign session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send an email to your Lotus Lead Project Manager withdrawing consent, and in the body of such request you must state your e-mail, full name, US Postal Address, and telephone number.

Required hardware and software

| Acquired nardware and software | |
|---|---|
| Operating Systems: | Windows® 2000, Windows® XP, Windows |
| | Vista® Mac OS® X |
| Browsers: | Final release versions of Internet Explorer® 6.0 |
| | or above (Windows only); Mozilla Firefox 2.0 |
| | or above (Windows and Mac); Safari <sup>TM</sup> 3.0 or |
| | above (Mac only) |
| PDF Reader: | Acrobat® or similar software may be required |
| | to view and print PDF files |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | Allow per session cookies |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, you will be asked to re-accept the disclosure. Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

# Acknowledging your access and consent to receive materials electronically

By checking the "I agree to use Electronic Records and Signatures" box in the DocuSign system, you are confirming to us that:

- You can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC CONSUMER DISCLOSURES document; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify Lotus Clinical Research, LLC, as described above, you consent to receive through electronic means documents that require your signature